CLINICAL TRIAL: NCT07303335
Title: Prevalence of Sarcopenia in Patients Admitted to ICU and Its Progression During Hospitalization.
Acronym: SARC-ICU
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: P/25-054/Fundació assistencial; Mutua Terrassa (Other: Fundació Assistencial Mutua Terrassa)
Record Dates: First submitted 2025-11-17; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia; Critical Illness; Intensive Care (ICU) Myopathy; Body Composition Measurement; Bio-Impedance Measurements; Ultrasound Evaluation
MeSH Terms: conditions — Sarcopenia; Critical Illness; Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill adults (medical or surgical) expected to require prolonged mechanical ventilation.: Assesment of the body composition using Rectus Femoris (RF) Ultrasound and Bioelectrical Impedance Analysis (BIA)

SUMMARY:
This is a prospective, observational study at the ICU of Hospital Mútua de Terrassa, running from May to December 2025. The primary goal is to determine the prevalence of sarcopenia in adult patients requiring more than 48 hours of mechanical ventilation. Sarcopenia is assessed using the SARC-F score, impedanciometry, and quadriceps ultrasound. Secondary aims include tracking the development of ICU-Acquired Weakness (ICU-AW) using the MRC score. All data is collected anonymously after obtaining informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old.
* Expected duration of mechanical ventilation (MV) exceeding 48 hours.

Exclusion Criteria:

* Refusal to participate.
* Mechanical ventilation not exceeding 48 hours.
* Do-not-resuscitate (DNR) orders or limitations of therapeutic effort upon admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a polyvalent (medical and surgical) ICU.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sarcopenia at the time of ICU admission. | Baseline at admission to ICU
  Describe the prevalence of sarcopenia at the time of ICU admission in patients with an expected duration of mechanical ventilation (MV) exceeding 48 hours.

SECONDARY OUTCOMES:
Detecting patients who develop ICU-Acquired Weakness (ICU-AW) and/or prolonged mechanical ventilation weaning | From ICU admission to 30 days follow-up
  Detecting patients who develop ICU-Acquired Weakness (ICU-AW) and/or prolonged mechanical ventilation weaning, defined as failure of definitive disconnection from mechanical ventilation
Detecting the appearance of other complications | From admission to 30 days follow up
  Detecting the appearance of other complications during admission such as: the appearance of refeeding syndrome or increased prevalence of insulin resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Mútua Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Sostakaite G, Jauniskyte M, Budrys D, Budrevicius K, Salciute-Simene E, Svetikiene M, Jovaisa T, Zvirblis T, Klimasauskas A, Sipylaite J. Comparison of Two Techniques to Assess Muscle Mass Loss During ICU Stay: Muscle Ultrasound vs Bioelectrical Impedance Analysis. Nutrition. 2025 Feb;130:112607. doi: 10.1016/j.nut.2024.112607. Epub 2024 Oct 24. PMID 39549651
- [Background] Nakanishi N, Tsutsumi R, Okayama Y, Takashima T, Ueno Y, Itagaki T, Tsutsumi Y, Sakaue H, Oto J. Monitoring of muscle mass in critically ill patients: comparison of ultrasound and two bioelectrical impedance analysis devices. J Intensive Care. 2019 Dec 16;7:61. doi: 10.1186/s40560-019-0416-y. eCollection 2019. PMID 31890223

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT07303335/Prot_SAP_000.pdf